CLINICAL TRIAL: NCT06926491
Title: A Multicenter, Open-label, Single-arm, Phase 3 Study of KK8398 (Infigratinib) in Patients With Achondroplasia (AOBA Study)
Brief Title: Evaluate the Efficacy and Safety of KK8398 in Patients With Achondroplasia（AOBA Study）
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8398-001; jRCT2031240562 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2025-04-01; First posted 2025-04-13 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Achondroplasia
MeSH Terms: conditions — Achondroplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KK8398 (Experimental)
  Interventions: Drug: KK8398

INTERVENTIONS:
Drug: KK8398 — KK8398 will be administered.

SUMMARY:
This trial will evaluate the efficacy of KK8398 on annualized height velocity after 52 weeks of repeated administration of KK8398 to patients with achondroplasia

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are between 2.5 and 17.5 years old of age at the time of provisional registration. Patients who meet certain criteria in terms of Tanner stage and bone age.
2. Patients who have been diagnosed with achondroplasia through genetic testing.

Exclusion Criteria:

1. Patients who meet the criteria for a certain height determined by age and gender in the "Growth Chart for Patients with Achondroplasia" at the time of the pre-registration examination
2. Patients who have received treatment with r-hGH or a CNP analogue within a certain period prior to the pre-enrollment examination.
3. Patients who have had previous osteotomy or who are scheduled to undergo osteotomy or epiphyseal growth inhibition during the study period. Epiphyseal growth inhibition in which the plate was removed more than 26 weeks prior to the pre-registration examination will not be excluded if the patient has completely healed without sequelae, based on the judgment of the investigator or sub-investigator.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2031-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in annualized height velocity | Pre-dose, Week 52

SECONDARY OUTCOMES:
Height Z-score using growth tables in patients with achondroplasia and the change from baseline | Pre-dose, Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Yu Sato, Study Director — Kyowa Kirin Co., Ltd.
Locations (9):
- Japan (9):
  - Aichi Children's Health and Medical Center, Ōbu, Aichi-ken
  - Osaka University Hospital, Suita, Osaka
  - Osaka Women's and Children's Hospital, Waizumi, Osaka
  - Tokyo Metropolitan Children's Medical Center, Fuchū, Tokyo
  - Tottori University Hospital, Yonago, Tottori
  - Niigata University Medical and Dental Hospital, Niigata
  - Okayama University Hospital, Okayama
  - ISEIKAI International General Hospital, Osaka
  - Osaka City General Hospital, Osaka

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.